CLINICAL TRIAL: NCT03559374
Title: Study of Vanadis® NIPT for Non-invasive Prenatal Screening of Trisomies (T21, T18 and T13)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: PerkinElmer, Wallac Oy (Industry)
Collaborators: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Sponsor
Other Study IDs: F01-16013
Record Dates: First submitted 2018-05-17; First posted 2018-06-18 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Trisomy 21; Trisomy 18; Trisomy 13
Keywords: Vanadis NIPT system
MeSH Terms: conditions — Down Syndrome; Trisomy 18 Syndrome; Trisomy 13 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Consenting women will provide samples to be tested with Vanadis NIPT system.
  Interventions: Other: Vanadis NIPT system

INTERVENTIONS:
Other: Vanadis NIPT system — A novel cost effective not NGS (next-generation sequencing) test, based on imaging single DNA molecules for high precision NIPT (non-invasive prenatal testing)

SUMMARY:
This study will assess the feasibility of Vanadis NIPT for screening of T21, T18 and T13. The results obtained from Vanadis NIPT will be compared with the study site's current prenatal screening methods. The primary objectives are: 1) To assess the feasibility of Vanadis NIPT for screening of T21, T18 and T13 in the maternal healthcare setting, 2) To assess preliminary performance of Vanadis NIPT for screening of T21 in comparison to site's routine screening methods i.e. combined and integrated tests, and 3) To evaluate preliminary cost effectiveness of Vanadis NIPT use in different models. The secondary objective is to assess the feasibility of Vanadis NIPT regarding determination of fetal sex.

ELIGIBILITY:
Inclusion Criteria:

* between the age of 18 and 55 years (inclusive)
* ≥ 10+0 weeks gestation

Exclusion Criteria:

* Pregnant woman undergoing amniocentesis without any screening test result
* Pregnant woman with previous severe hypotension episodes or other conditions that may complicate the blood sampling
* Known maternal aneuploidy
* Known maternal cancer
* Invasive test (chorionic villus sampling or amniocentesis) performed before blood sampling for NIPT

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 1. Pregnant women attending the clinic for chorionic villus sampling or amniocentesis and have combined or integrated screening test result available
  2. Pregnant women attending the clinic for chorionic villus sampling and willing to have combined or integrated screening test result for study purposes
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Assess preliminary performance of Vanadis NIPT for screening of T21 in comparison to site's routine screening methods i.e. combined and integrated tests | Three weeks

SECONDARY OUTCOMES:
Assess the feasibility of Vanadis NIPT for screening of T21, T18 and T13 in comparison to fetal karyotype from invasive testing, and by evaluating overall usability of the test in routine laboratory work. | Three weeks
  Evaluation includes the follow up for each woman and matching the results of combined and integrated test and with the results of NIPT and karyotype. Feasibility will be assessed by determining the concordance between chromosomal abnormalities determined by Vanadis NIPT and trisomies confirmed by karyotype analysis, and by assessing the overall usability in the public healthcare setting by evaluating e.g. turnaround time and user friendliness.
Evaluate preliminary cost effectiveness of Vanadis NIPT by evaluating resources, false positive rates and detection rates | Three weeks
  Cost effectiveness will be evaluated when the test is offered to all women or only women with T21 risk between 1:100 and 1:2500 or between 1:11 and 1:1000, or alternatively to 3000 or 10000 women annually. Cost effectiveness will be assessed by taking into account the costs of NIPT, combined test, invasive procedure, fetal karyotype and counselling, the potential benefits (rate of reduction of invasive procedures, miscarriages, births with trisomy 21) and births with chromosomal diseases undetectable with NIPT.
Assess feasibility of Vanadis NIPT regarding determination of fetal sex by comparing the Vanadis NIPT result with the fetal karyotype from invasive testing | Three weeks

CONTACTS AND LOCATIONS:
Overall Officials: Enza Pavanello, Principal Investigator — Centro Screening neonatale e prenatale del Piemonte e Valle d'Aosta AOU Città della Salute e della Scienza di Torino
Locations (1):
- Centro Screening neonatale e prenatale del Piemonte e Valle d'Aosta AOU Città della Salute e della Scienza di Torino, Turin, Italy

IPD SHARING:
Plan to Share IPD: No